CLINICAL TRIAL: NCT03673475
Title: Internal Jugular Vein Distensibility and Pleth Variability Index for Evaluating Fluid Responsiveness
Brief Title: Internal Jugular Vein Distensibility and Pleth Variability Index(PVI) for Evaluating Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, MELTEM CAKMAK, Anesthesiologist, Tepecik Training and Research Hospital
Other Study IDs: Meltem Cakmak
Record Dates: First submitted 2018-08-24; First posted 2018-09-17 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Intravascular Volume

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fluid responsiveness: Assessment of fluid responsiveness using pleth variebility index and jugular vein distensibility in patients undergoing major abdominal surgery
  Interventions: Procedure: Assessment of fluid responsiveness

INTERVENTIONS:
Procedure: Assessment of fluid responsiveness — assessment of intravascular volume status using pleth variebility index and internal jugular vein distensibility in major abdominal surgery

SUMMARY:
Assessment of intravascular volume status is crucial in order to predict the efficacy of volume status in major abdominal surgery. The aim of the study is to verify the feasibility and usefulness of the internal jugular vein distensibility index as an adjunct to the pleth variebility index(PVI) to predict fluid responsiveness in major abdominal surgery.

DETAILED DESCRIPTION:
Forty patients above age 18 and ASA status I-III who are undergoing major abdominal surgery will be enrolled in the study. patients with right heart failure, arrythmia, severe valve stenosis or regurgitation will be excluded. After induction of general anesthesia, when the patients are hemodynamically stabilised, PVI and jugular vein distensibility will be calculated and recorded. after volume load with 500 ml gel infusion(in 15 min), measurements will be repeated within 10 minutes and recorded. Patients will be allocated to 2 groups according to the change in mean arterial pressure(MAP) after volume expansion: Responders will be defined as an increase in MAP by >%10; while nonresponders will be defined as an increase in MAP <%10 or decrease in MAP.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists(ASA) physical status I-III patients
* patients undergoing major abdominal surgery

Exclusion Criteria:

* arrythmia
* severe right ventricle failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
number of patients with significant change in VJI distensibility and pleth variebility index | during surgery at day 0
  volume responders with significant change in jugular vein distensibility and pleth variebility index

CONTACTS AND LOCATIONS:
Overall Officials: Yucel Karaman, ass. prof, Study Chair — Tepecik TRH
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No